CLINICAL TRIAL: NCT00913432
Title: A 12-week With Possible Extension, Prospective, Multicenter, Randomized, Open Label, Uncontrolled, 2-parallel Group, Phase II Study to Compare Efficacy and Safety of AB1010 at 3 and 6 mg/kg/Day in Combination With Methotrexate, in Treatment of Patients With Active Rheumatoid Arthritis With Inadequate Response to 1. Methotrexate or to 2. Any DMARD Including Anti TNF Alpha if Patients Previously Failed Methotrexate or to 3. Methotrexate in Combination With Any DMARD Including Anti TNF Alpha
Brief Title: Masitinib in Combination With Methotrexate, in Treatment of Patients With Active Rheumatoid Arthritis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: AB Science (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: AB06010
Record Dates: First submitted 2009-06-03; First posted 2009-06-04 (Estimated); Last update posted 2018-12-13 (Actual); Status verified 2018-12

CONDITIONS: Rheumatoid Arthritis
Keywords: rheumatoid arthritis; methotrexate; DMARD; c-kit inhibitor
MeSH Terms: conditions — Arthritis, Rheumatoid | interventions — masitinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- masitinib 3 mg (Experimental): masitinib 3 mg/kg/day
  Interventions: Drug: masitinib
- masitinib 6 mg (Experimental): masitinib 6 mg/kg/day
  Interventions: Drug: masitinib

INTERVENTIONS:
Drug: masitinib — 3 mg/kg/day oral route
  Other Names: AB1010
  Arms: masitinib 3 mg
Drug: masitinib — masitinib 6 mg/kg/day oral route
  Other Names: AB1010
  Arms: masitinib 6 mg

SUMMARY:
A 12-week with possible extension, phase II study to compare efficacy and safety of masitinib at 3 and 6 mg/kg/day in combination with methotrexate, in treatment of patients with active rheumatoid arthritis refractory to standard treatments.

ELIGIBILITY:
Inclusion Criteria:

1. Disease duration of at least 6 months Meet American College of Rheumatology (ACR) criteria for RA.
2. ACR functional class I-III
3. Have active RA
4. Failed (defined as active RA with stable dose during 3 months) i. methotrexate or ii. any DMARD including anti TNF alpha if patients previously failed methotrexate or iii. methotrexate in combination with any DMARD including anti TNF alpha

Exclusion Criteria:

1. Patient had a major surgery within 2 weeks prior to study entry.
2. Life expectancy < 6 months.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2007-03; Primary Completion 2009-06 (Actual); Study Completion 2010-09 (Actual)

PRIMARY OUTCOMES:
American College of Rheumatology Score 50 | week 12

SECONDARY OUTCOMES:
DAS28 | week 4, 8 and 12

CONTACTS AND LOCATIONS:
Overall Officials: Jacques Tebib, MD, PhD, Principal Investigator — CHU de Lyon Sud